CLINICAL TRIAL: NCT04789213
Title: Comparison of Mortality, Morbidity and Risk Factors in Living- Donor and Deceased-Donor Liver Retransplantation
Brief Title: Mortality, Morbidity and Risk Factors of Liver Retransplantation
Status: Completed | Type: Observational
Sponsor: Memorial Bahçelievler Hospital (Other)
Responsible Party: Principal Investigator, Kamil Yalçın Polat, Prof.Dr., Memorial Bahçelievler Hospital
Other Study IDs: MemorialBahcelievler1
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-12

CONDITIONS: Liver Transplant; Complications; Liver Transplant Rejection; Liver Transplant Failure; Liver Diseases; Liver Cirrhosis; Liver Failure; Organ Transplant Failure or Rejection
MeSH Terms: conditions — Liver Diseases; Liver Cirrhosis; Liver Failure; Rejection, Psychology | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Living Donor Liver Transplantation
  Interventions: Other: Liver Transplantation
- Patients with Deceased Donor Liver Transplantation
  Interventions: Other: Liver Transplantation

INTERVENTIONS:
Other: Liver Transplantation — Liver Transplantation

SUMMARY:
This study aims to compare the short and long term outcomes of living donor and deceased donor liver retransplantation. Bearing that in mind, the investigators will retrospectively analyze the files of patients whom underwent a liver retransplantation in Memorial Bahcelievler Hospital Organ Transplantation Center.

ELIGIBILITY:
Inclusion Criteria:

* Having a liver retransplantation

Exclusion Criteria:

* N/A

Min Age: 0 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with liver failure who underwent a second liver transplantation (i.e. re-transplantation)
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Survival ratio | 1 minutes
  Overall graft and patient survival ratio

SECONDARY OUTCOMES:
Morbidity | 10 minutes
  Postoperative complications such as septicemia, hepatic artery thrombosis etc.
Peri-operative informations | 15 minutes
  Peri-operative informations such as blood loss during surgery
Blood Test Results | 20 minutes
  Patients' blood test results specific to liver such as International Normalization Ratio

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Yalçın Polat, Prof, Principal Investigator — Memorial Bahçelievler Hospital
Locations (1):
- Memorial Bahçelievler Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No